CLINICAL TRIAL: NCT03475472
Title: Direct Molecular Characterization of Bacteria From Tracheal and Urine Samples in Patients Hospitalized at the Intensive Care Units at the University Hospital of Basel and at the REHAB Basel
Brief Title: Direct Molecular Characterization of Bacteria From ICU and From the REHAB
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00049; me17Khanna2
Record Dates: First submitted 2018-02-14; First posted 2018-03-23 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bacteria from tracheal and urinary samples routinely taken in intensive care units (ICU) and REHAB-Basel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators aim to directly investigate the molecular properties of bacteria from tracheal and urinary samples routinely taken in intensive care units (ICU) patients.

DETAILED DESCRIPTION:
Investigators goal is to determine major bacterial activities and properties in the infected patient as a basis for more targeted, efficient antimicrobial discovery. Investigators will determine the abundance of dozens to hundreds of pathogen proteins in the samples and in in vitro cultures of the same pathogen strains using cutting-edge ultra-sensitive proteomics approaches (Parallel reaction Monitoring (PRM), Sequential Windowed Acquisition of All Theoretical Fragment Ion Mass Spectra (SWATH-MS). Data will be analyzed using dedicated mass spectrometry and proteomics packages using parametric and non-parametric statistics (false discovery rate determination based on decoy databases; t-tests of log-transformed abundance data with Benjamin-Hochberg corrections for multiple testing, normal distribution of the data will be evaluated by Kolmogorov-Smirnov test).

Based on experience from in vitro and animal infection experiments, a sample size of 10 can reveal 2fold differences in protein abundance among 500 top proteins at a significance of α = 0.05 and a power of β = 0.8 (after correction for multiple testing). However, it is possible that human patient samples have higher variance compared to animal infection models. Investigators will thus use a sequential statistics approach in which they continuously adjust sample size estimates based on the variance of the accumulating data. It may be possible that no sufficient sample sizes for all bacterial pathogens of interest will be reached within two years.

ELIGIBILITY:
Inclusion Criteria:

* confirmed infection of lung or urine by one or several members of a defined set of bacterial pathogens (Pseudomonas aeruginosa, E. coli, Klebsiella spp., Serratia marcescens, Enterobacter spp., Acinetobacter baumannii, Staphylococcus aureus, Streptococcus pneumonia

Exclusion Criteria:

* Proof of a refusal to the general research consent
* No detected bacteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All in ICU-patients and REHAB-Basel patients with residual material from tracheal or urinary samples taken for routine diagnostics of patients with suspected bacterial infection will be included.
Sampling Method: Probability Sample
Enrollment: 971 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Abundance of pathogen proteins | once during study (February 2018 until June 2020) but no fixed timepoint
  Determine the abundance of pathogen proteins in the samples and in in vitro cultures of the same pathogen strains using cutting-edge ultra-sensitive proteomics approaches (Parallel reaction monitoring, PRM, Sequential Windowed Acquisition of All Theoretical Fragment Ion Mass Spectra, SWATH-MS). Data will be analyzed using dedicated mass spectrometry and proteomics packages using parametric and non-parametric statistics (false discovery rate determination based on decoy databases; t-tests of log-transformed abundance data with Benjamin-Hochberg corrections for multiple testing, normal distribution of the data will be evaluated by Kolmogorov-Smirnov test).

CONTACTS AND LOCATIONS:
Overall Officials: Nina Khanna, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - Division of Infectious Diseas and Hospital Epidemiology, Basel
  - REHAB Basel, Klinik für Neurorehabilitation und Paraplegiologie, Basel